CLINICAL TRIAL: NCT00030758
Title: G-CSF (Filgrastim) or Pegfilgrastim Secondary Prophylaxis In The Adjuvant Chemotherapy Of Early Breast Cancer
Brief Title: Filgrastim or Pegfilgrastim in Preventing Neutropenia in Women Receiving Chemotherapy Following Surgery for Breast Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Anglo Celtic Cooperative Oncology Group (Other)
Collaborators: Scottish Cancer Therapy Network (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: ACCOG-SCTN-BR0101; CDR0000069195 (Registry Identifier: PDQ (Physician Data Query)); SCTN-BR0101; EU-20143
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2007-06

CONDITIONS: Breast Cancer; Neutropenia
Keywords: neutropenia; stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neutropenia | interventions — Filgrastim; pegfilgrastim

INTERVENTIONS:
Biological: filgrastim
Biological: pegfilgrastim

SUMMARY:
RATIONALE: Colony-stimulating factors, such as filgrastim or pegfilgrastim, may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy. It is not yet known whether filgrastim or pegfilgrastim is more effective than standard treatment in preventing neutropenia in women who are receiving adjuvant chemotherapy for breast cancer.

PURPOSE: Randomized phase IV trial to compare the effectiveness of filgrastim or pegfilgrastim with that of standard treatment in preventing neutropenia in women who are receiving chemotherapy after undergoing surgery for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of filgrastim (G-CSF) or pegfilgrastim as secondary prophylaxis versus standard management after the first neutropenic event in maintaining dose-intensity of adjuvant chemotherapy in patients with early breast cancer.
* Determine the proportion of patients who experience at least one neutropenic event.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age (60 and under vs over 60) and participating center.

Patients receive chemotherapy as per local practice. After the first neutropenic event, patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive filgrastim (G-CSF) subcutaneously (SC) for 7 days beginning 2 days after the final dose in a course of adjuvant chemotherapy (e.g., beginning on day 3 for a course of chemotherapy administered on day 1 only OR beginning on day 10 for a course of chemotherapy administered on days 1 and 8) OR a single dose of pegfilgrastim SC administered approximately 24 hours after chemotherapy that is administered on day 1 only.
* Arm II: Patients receive standard conservative management. Patients are followed for up to 10 years.

PROJECTED ACCRUAL: A total of 400 patients will be accrued for this study within 7 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer

  * No locally advanced or metastatic breast cancer, including supraclavicular fossa metastases
* Prior neutropenic event on current chemotherapy regimen, defined as 1 of the following:

  * Hospitalization due to neutropenia
  * Absolute neutrophil count ≤ 1.5 times upper limit of normal and considered sufficiently low to require a treatment delay or a dose reduction > 15% of planned dose
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other concurrent malignancy
* Considered suitable risk and fitness status to continue adjuvant chemotherapy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior filgrastim (G-CSF) or pegfilgrastim

Chemotherapy:

* See Disease Characteristics
* No prior chemotherapy other than current regimen

Endocrine therapy:

* Prior tamoxifen allowed

Radiotherapy:

* Concurrent radiotherapy allowed
* No concurrent sandwich/synchronous radiotherapy (i.e., administered during a break in the chemotherapy regimen)

Surgery:

* See Disease Characteristics

Other:

* Concurrent enrollment on other licensed chemotherapy trials allowed provided G-CSF is not excluded (e.g., TACT or TANGO trials)
* Concurrent enrollment in the sequential arm of the SECRAB trial allowed (synchronous arm ineligible)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 816 (Estimated)
Dates: Start 2001-10

PRIMARY OUTCOMES:
Proportion of patients achieving ≥ 85% of planned dose intensity
Proportion of patients with ≥ 1 neutropenic event

SECONDARY OUTCOMES:
Dose intensity achieved
Cost of management

CONTACTS AND LOCATIONS:
Overall Officials: Robert C.F. Leonard, MD, BS, MB, Study Chair — Charing Cross Hospital; Kirsten Murray, Study Chair — Scottish Cancer Therapy Network
Locations (32):
- United Kingdom (32):
  - City Hospital - Birmingham, Birmingham, England
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Cheltenham General Hospital, Cheltenham, England
  - Princess Alexandra Hospital, Essex, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - King George Hospital, Ilford, Essex, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Queen Elizabeth Hospital NHS Trust, London, England
  - King's College Hospital, London, England
  - St. George's Hospital, London, England
  - Christie Hospital NHS Trust, Manchester, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - Northampton General Hospital NHS Trust, Northampton, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Royal Oldham Hospital, Oldham, England
  - Peterborough Hospitals Trust, Peterborough, England
  - Berkshire Cancer Centre at Royal Berkshire Hospital, Reading, England
  - Oldchurch Hospital, Romford, England
  - Salisbury District Hospital, Salisbury, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - South Tyneside District Hospital, South Shields, England
  - Southampton University Hospital NHS Trust, Southampton, England
  - Sunderland Royal Hospital, Sunderland, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - Yeovil District Hospital, Yeovil - Somerset, England
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Scottish Cancer Therapy Network, Edinburgh, Scotland
  - West of Scotland Cancer Centre, Glasgow, Scotland
  - Royal Infirmary - Castle, Glasgow, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Singleton Hospital of the Swansea NHS Trust, Swansea, Wales